CLINICAL TRIAL: NCT02499588
Title: Observational User Evaluation of the Peristomal Skin Condition in Ostomates Using ConvaTec Moldable Technology™
Brief Title: User Evaluation of the Peristomal Skin Condition in Ostomates Using ConvaTec Moldable Technology™
Acronym: OSMOSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-0509-15-U375
Record Dates: First submitted 2015-07-03; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Colostomy; Ileostomy; Urostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Esteem Plus with ConvaTec Moldable Technology
Device: Natura with ConvaTec Moldable Technology
Device: Natura Accordion with ConvaTec Moldable Technology
Device: Esteem synergy Plus with ConvaTec Moldable Technology

SUMMARY:
The primary aim of this study is to demonstrate the maintenance of healthy peri-stomal skin over a two month period in subjects who use ConvaTec Moldable Technology™ Skin Barriers as part of their standard protocol of care following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 years old and older.
* Subjects who agree to participate in the evaluation and who have signed the informed consent form.
* Subjects presenting with a stoma (ileostomy, colostomy or urostomy).
* Subjects for whom ConvaTec Moldable Technology™ per package insert, within the context of routine clinical care is used as the first long-term (within 7 days of ostomy surgery) system following surgery and who have intact peristomal skin (healthy or SACs L1).

Exclusion Criteria:

* Subjects who, according to the investigator, have cognitive problems that prevent them from answering a questionnaire or for whom the evaluation could be a problem.
* Subjects who are in a simultaneous clinical evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with colostomy, ileostomy or urostomy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Peri-stomal skin condition at 8-15 days following the application of the barrier. | 8-15 days
  Using SACs scale to determine incidence and severity of lesions

SECONDARY OUTCOMES:
Peristomal skin condition in ostomates at 1 month (± 15 days) following the application of the barrier. | 1 month (± 15 days)
  Using SACs scale to determine incidence and severity of lesions
Peristomal skin condition in ostomates at 2 months (± 15 days) following the application of the barrier. | 2 months (± 15 days)
  Using SACs scale to determine incidence and severity of lesions

CONTACTS AND LOCATIONS:
Overall Officials: Kim Peters, BSc (Hons), Study Director — Sponsor GmbH
Locations (1):
- Voivodeship Specialistic Hospital in Gorzow Wlkp., Gorzów Wielkopolski, Lubusz Voivodeship, Poland